CLINICAL TRIAL: NCT04795765
Title: Prospective SpineJack System Registry
Brief Title: SpineJack System Postmarket Registry
Status: Completed | Type: Observational
Sponsor: Stryker Instruments (Industry)
Collaborators: Talosix (Unknown)
Responsible Party: Sponsor
Other Study IDs: SISSJS2019US
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Osteoporotic Vertebral Compression Fractures
MeSH Terms: interventions — Kyphoplasty; Vertebroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients treated with SpineJack system: SpineJack system procedure
  Interventions: Procedure: SpineJack system
- Patients treated with vertebral augmentation: Vertebral augmentation procedures may include either balloon kyphoplasty (BKP) or vertebroplasty (VP).
  Interventions: Procedure: Balloon kyphoplasty; Procedure: Vertebroplasty

INTERVENTIONS:
Procedure: SpineJack system — For use in the reduction of painful osteoporotic vertebral compression fractures.
  Groups: Patients treated with SpineJack system
Procedure: Balloon kyphoplasty — Treatment of osteoporotic vertebral compression fractures.
  Groups: Patients treated with vertebral augmentation
Procedure: Vertebroplasty — Treatment of osteoporotic vertebral compression fractures.
  Groups: Patients treated with vertebral augmentation

SUMMARY:
This postmarket registry is intended to prospectively collect real world data to support ongoing safety and performance of the SpineJack system.

DETAILED DESCRIPTION:
The SpineJack System Registry will employ a prospective, multicenter, observational, consecutive enrollment design. The sample size for this Registry will include at least 400 patients treated for VCFs across approximately 10 sites. A total of 240 patients will be treated with the SpineJack system and 160 patients will be treated with other vertebral augmentation (VA) procedures, such as BKP or VP. Sites within the U.S. may include healthcare professionals (HCPs) that are surgeons, pain physicians and/or interventional radiologists.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Understand and sign the informed consent form (as applicable)
3. Exhibit no altered mental status or language barrier that may prevent completion of the patient reported outcome (PRO) surveys following the procedure.
4. VCF diagnosis made and/or confirmed at participating site.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients that meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Back pain | 12 months post-procedure
  The numeric rating scale consists of an eleven-point scale used for patient self-reporting of back pain, which ranges from 0 (no pain) to 10 (the worst pain imaginable).
Radiological outcomes | Immeditely post-procedure
  Vertebral body height restoration
Radiological outcomes | Immediately post-procedure
  Adjacent level fractures
Adverse events | 12 months post-procedure
  1. Incidence of adverse device effects (ADEs) and serious adverse device effects (SADEs) requiring surgical re-intervention or re-treatment at the treated level
  2. Incidence of unanticipated ADEs
  3. Incidence of procedure-related AEs
Quality of life indices - Roland Morris Disability Questionnaire (RMDQ) | 12 months post-procedure
  24-item self-report questionnaire used in patients with mild to moderate disability due to acute, sub-acute or chronic low back pain
Patient-Reported Outcomes Measurement Information System (PROMIS Global-10) | 12 months post-procedure
  10-item questionnaire that is used to assess general domains of health and functioning, including overall physical health, mental health, social health, pain, fatigue and overall perceived quality of life

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - San Diego Neurosurgery, Encinitas, California
  - California Orthopedics and Spine, Larkspur, California
  - Cleveland Clinic, Stuart, Florida
  - St. Luke's IntermountainResearch Center, Boise, Idaho
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Clinical Investigations, Edmond, Oklahoma
  - Center for Diagnostic Imaging (CDI), Puyallup, Washington
  - Rainier Orthopedic Institute, Puyallup, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin